CLINICAL TRIAL: NCT03383237
Title: Clinical Study of Apatinib as the Second-line Therapy in Malignant Melanoma：An Open-Label, Single-center, Single-arm Study
Brief Title: Clinical Study of Apatinib as the Second-line Therapy in Malignant Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP051
Record Dates: First submitted 2017-12-18; First posted 2017-12-26 (Actual); Last update posted 2017-12-27 (Actual); Status verified 2017-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): Apatinib 500mg/d,q.d.,p.o.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500mg/d,q.d.,p.o.

SUMMARY:
The purpose of this study is to confirm the safety and efficacy of Apatinib as the Second-line Therapy in Malignant Melanoma.

DETAILED DESCRIPTION:
Melanoma is a malignant tumor caused by hyperplasia of abnormal melanoma cells.Most of the adults above 30 years of age occur in the skin, mucosa and internal organs. The investigators designed the study to explore the possibility of apatinib as the Second-line Therapy in Malignant Melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form prior to patient entry.
2. Pathologically confirmed first-line treatment of advanced malignant melanoma patients with at least one measurable lesion.
3. ≥ 18 and ≤ 70 years of age.
4. Eastern Cooperative Oncology Group(ECOG) performance status 0 or 1.
5. Life expectancy of more than 3 months.
6. Adequate hepatic, renal, heart, and hematologic functions: ANC ≥ 1.5×109/L, PLT ≥ 100×109/L, HB ≥ 90 g/L, TBIL ≤ 1.5×ULN, ALT or AST ≤ 2.5×ULN (or ≤ 5×ULN in patients with liver metastases), Serum Cr ≤ 1.5×ULN, Cr clearance ≥ 60 mL/min;Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (50%).
7. Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 6 months after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 6 months after last dose of study drug.

Exclusion Criteria:

1. uncontrollable hypertension (systolic BP ≥140 mmHg or diastolic BP ≥90 mmHg, despite optimal medical therapy), grade II The above myocardial ischemia or myocardial infarction, poor control of arrhythmia (including QTc interval male ≥ 450 ms, female ≥ 470 ms).
2. Patients previously treated with anticancer therapies also have a Toxicity Level> 1 in NCI CTCAE.
3. A variety of factors that affect oral absorption (such as inability to swallow, nausea, vomiting, chronic diarrhea, intestinal obstruction, etc.).
4. Patients with gastrointestinal bleeding risk may not be included, including the following: (1) active peptic ulcer lesions and fecal occult blood (++); (2) history of melena and vomiting within 3 months; (3) ) For fecal occult blood (+) must be gastroscopy, clear whether the existence of gastrointestinal organic diseases.
5. Coagulation dysfunction (INR> 1.5, PT> ULN + 4s or APTT> 1.5 ULN), with bleeding tendency or ongoing thrombolysis or anti-blood coagulation treatment.
6. Long-term, unhealed wounds or fractures.
7. Active bleeding, within 30 days after major surgery.
8. Intracranial metastasis.
9. Pregnant or lactating women.
10. Cytotoxic drug treatment, radiotherapy within 3 weeks after treatment; had taken two or more targeted drugs, or into the group before the other three months have been taking other targeted drugs.
11. Other malignant tumors in the past 3 years.
12. The investigators believe there is any condition that may harm the subject or result in the subject's inability to meet or perform the research requirements.
13. Huge metastasis / recurrence (tumor diameter> 5 cm)。
14. Malignant pleural effusion or ascites, causing NCI CTCAE grading 2 or more people with dyspnea.
15. Any allergy to apatinib should be excluded.
16. Severe liver and kidney dysfunction (grade 4) patients should be excluded.
17. Persons with a history of substance abuse who can not be abdicated or have mental disorders.
18. According to the judgment of the researcher, there is a concomitant disease that seriously endangers the patient's safety or affects the patient in completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | up to 2 year
  From date of randomization until the date of first documented progression or date of death from any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 1 year
  From date of randomization until the date of death from any cause
Disease Control Rate (DCR) | up to 1 year
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Overall survival(OS) | up to 2 year
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zibing Wang, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Yuan S, Fu Q, Zhao L, Fu X, Li T, Han L, Qin P, Ren Y, Huo M, Li Z, Lu C, Yuan L, Gao Q, Wang Z. Efficacy and Safety of Apatinib in Patients with Recurrent or Refractory Melanoma. Oncologist. 2022 Jun 8;27(6):e463-e470. doi: 10.1093/oncolo/oyab068. Erratum In: Oncologist. 2022 Aug 5;27(8):e684. doi: 10.1093/oncolo/oyac103. PMID 35348754